CLINICAL TRIAL: NCT07040826
Title: Pharmacokinetics and Safety Study of Lifitegrast Eye Drops in Healthy Subjects - A Single-Center, Randomized, Double-Blind, Single-Dose, Two-Period Crossover Design Phase I Clinical Trial
Brief Title: Lifitegrast Eye Drops in Healthy Subjects：Phase I Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL-YJ1-039-101
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifitegrast (T) on Day 1, then Xiidra® (R) on Day 8. (Experimental)
  Interventions: Drug: Xiidra
- Xiidra® (R) on Day 1, then Lifitegrast (T) on Day 8. (Experimental)
  Interventions: Drug: Lifitegrast

INTERVENTIONS:
Drug: Xiidra — Administered on Day 1 to subjects in Group B, and on Day 8 to subjects in Group A as part of a crossover study design.
  Arms: Lifitegrast (T) on Day 1, then Xiidra® (R) on Day 8.
Drug: Lifitegrast — Administered on Day 1 to subjects in Group A, and on Day 8 to subjects in Group B as part of a crossover study design.
  Arms: Xiidra® (R) on Day 1, then Lifitegrast (T) on Day 8.

SUMMARY:
This is a single-center, randomized, double-blind, single-dose, two-period crossover Phase I clinical trial designed to:

* Compare the pharmacokinetic (PK) profiles of Lifitegrast Ophthalmic Solution and Xiidra® in plasma and tears following single-dose administration in healthy subjects.
* Evaluate the safety and tolerability of Lifitegrast Ophthalmic Solution in healthy subjects.

A total of 24 healthy subjects will be randomized into two treatment sequences (Group A: T/R; Group B: R/T). The study duration per subject will be approximately 36 days, including:

* Screening Period (Day -21 to Day -1)
* Treatment Periods (Day 1, followed by a 7-day washout period, then Day 8 or early termination)
* Safety Follow-up (Day 15, 7 days after the last dose).

On Day 1 of Cycle 1, one study eye will be selected and designated for all subsequent tear PK sampling. Treatment assignments:

* Group A: Lifitegrast (T) on Day 1, then Xiidra® (R) on Day 8.
* Group B: Xiidra® (R) on Day 1, then Lifitegrast (T) on Day 8. Each subject will receive one drop of the assigned medication (either Lifitegrast or Xiidra®) in each eye from the same single-dose container. Blood and tear samples will be collected per protocol for PK analysis, including parameters such as Cmax, AUC0-∞, AUC0-t, Tmax, T1/2, λz, and AUC_%Extrap. The PK profiles between the two treatments will be compared to evaluate bioequivalence and assess the safety of Lifitegrast Ophthalmic Solution.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the following criteria to be eligible:
* Healthy, aged 18-50 (inclusive), all genders.
* Signed informed consent pre-screening; comprehension of study and ability to complete it per protocol.
* BMI 19-27 kg/m² (inclusive); ≥45 kg for females, ≥50 kg for males.
* Bilateral best-corrected visual acuity ≥4.7 (5m, 5-point logMAR).
* No reported eye discomfort/abnormalities 1 month before randomization.
* No history of dry eye disease, as assessed by the investigator.
* No history of ocular inflammation (e.g., allergic conjunctivitis, uveitis) per investigator judgment.
* Use effective contraception during study and 30 days post-last dose:

Females: non-pregnant, non-lactating; premenopausal use approved methods, no egg donation.

Males with fertile partners: vasectomy (≥30 days, no viable sperm) or approved contraception, no sperm donation.

* Non-smoker, remain smoke-free during study.
* No excessive alcohol (>14 units/week) or illicit drug use history; abstain from both during study.

Exclusion Criteria:

* Subjects will be excluded if they meet any of the following:
* History or current diseases/conditions (e.g., circulatory, endocrine disorders) that pose risks or interfere with the study, as judged by the investigator.
* Blood donation or loss >300 mL within 56 days before randomization; no blood donation during the study.
* Allergy to study medications (e.g., lifitegrast, excipients).
* Prior participation in non - placebo lifitegrast clinical trials.
* Clinically significant abnormal test results:

Vital signs: ear temp >37.7℃ or <35.4℃; pulse >100 or <60 bpm; systolic BP ≥150 or <90 mmHg; diastolic BP ≥90 or <50 mmHg.

ECG: QTcF ≥450 ms (male), ≥460 ms (female). Lab tests: abnormal blood/urine, coagulation, infectious markers, drug/alcohol screenings.

Abnormal abdominal ultrasound or eye exams.

* Intraocular/laser eye surgery within 12 months, other eye surgeries within 3 months before screening, or planned eye surgery during the study.
* Use of ophthalmic drugs (incl. artificial tears), anticholinergics, oral/nasal steroids within 1 month before screening or during the study.
* Tobacco/nicotine use within 6 months before randomization.
* Contact lens use within 1 month before randomization or during the study.
* Prescription/OTC/herbal medications within 2 weeks or 5 half - lives (longer) before randomization or during the study.
* Pregnancy, lactation, or positive pregnancy test at screening.
* Participation in drug/device trials within 30 days or 5 half - lives (longer) before screening, or planned participation during the study affecting results.
* Conditions increasing risks, affecting compliance, or deemed unsuitable by the investigator (e.g., needle phobia).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Day 1 & Day 8: Pre-dose, 10, 20, 30, 45 minutes, and 1 hour post-administration.
  Evaluated in plasma and tears.
Area Under the Plasma Concentration-Time Curve (AUC0-∞) | Day 1 & Day 8: Pre-dose, 10, 20, 30, 45 minutes, and 1 hour post-administration.
  Evaluated in plasma and tears.
Area Under the Plasma Concentration-Time Curve (AUC0-t) | Day 1 & Day 8: Pre-dose, 10, 20, 30, 45 minutes, and 1 hour post-administration.
  Evaluated in plasma and tears.
Time to Peak Plasma Concentration (Tmax) | Day 1 & Day 8: Pre-dose, 10, 20, 30, 45 minutes, and 1 hour post-administration.
  Assessment: Evaluated in plasma and tears.
5. Terminal Phase Half-Life (T1/2) | Day 1 & Day 8: Pre-dose, 10, 20, 30, 45 minutes, and 1 hour post-administration.
  Evaluated in plasma and tears
Elimination Rate Constant (λz) | Day 1 & Day 8: Pre-dose, 10, 20, 30, 45 minutes, and 1 hour post-administration.
  Evaluated in plasma and tears.
Percentage Extrapolated AUC (AUC_%Extrap) | Day 1 & Day 8: Pre-dose, 10, 20, 30, 45 minutes, and 1 hour post-administration
  Evaluated in plasma and tears.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, China